CLINICAL TRIAL: NCT01769716
Title: Umbilical Cord Blood Therapy for Children With Global Developmental Delay
Brief Title: Umbilical Cord Blood Therapy for Global Developmental Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MinYoung Kim, M.D. (Other)
Collaborators: CHA University (Other)
Responsible Party: Sponsor-Investigator, MinYoung Kim, M.D., Associate Professor, Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCBGDD
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Global Developmental Delay
Keywords: Global developmental delay; Umbilical cord blood; Rehabilitation
MeSH Terms: conditions — Learning Disabilities | interventions — Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: allogeneic cord blood transplantation for children with developmental delay
Oversight: Data Monitoring Committee: No

ARMS (1):
- Umbilical cord blood transplantation (Experimental): Allogeneic umbilical cord blood will be administered intravenously or intraarterially under non-myeloablative immunosuppression. In case of autologous umbilical cord blood, immunosuppression is not required.
  Interventions: Procedure: Umbilical cord blood transplantation

INTERVENTIONS:
Procedure: Umbilical cord blood transplantation
  Other Names: Autologous or Allogeneic Umbilical Cord Blood

SUMMARY:
This open-label study aims to evaluate the safety and efficacy of autologous or allogeneic umbilical cord blood therapy for children with global developmental delay.

DETAILED DESCRIPTION:
Global developmental delay is defined as significant delay in two or more of the following developmental domains: gross/fine motor, speech/language, cognition, social/personal, and activities of daily living.

Umbilical cord blood has been used for inherited metabolic diseases that feature global developmental delay and many experimental animal studies have revealed umbilical cord blood is useful to repair neurological impairments in brain.

ELIGIBILITY:
Inclusion Criteria:

* Global developmental delay
* Willing to comply with all study procedure

Exclusion Criteria:

* Medical instability including pneumonia or renal function at enrollment
* Poor cooperation of guardian,including inactive attitude for rehabilitation and visits for follow-up
* Uncontrolled persistent epilepsy
* Not eligible according to the principal investigator

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2012-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in Cognition | Baseline - 6 months - 12 months
  Korean Wechsler Preschool and Primary Scale of Intelligence (K-WPPSI) (Higher value means better cognitive function (K-WPPSI: below 70 - worst, over 130 - best)
Changes in Cognitive Neurodevelopmental Outcome | Baseline - 1 month - 3 months - 6 months - 12 months
  Korean version of Bayley Scale of Infant Development-II Mental Scales (Higher value means better cognitive function: raw score 0 - worst, 178 - best.)

SECONDARY OUTCOMES:
Changes in Motor Performance | Baseline - 1 month - 3 months - 6 months - 12 months
  GMPM (Gross Motor Performance Measure) as a standardized measurement tool for assessing quality of movement regarding 3 properties of 5 ones; alignment, coordination, dissociated movement, stability, and weight shift (range: 0~100, Higher value means better motor quality.)
Changes in Standardized Gross Motor Function | Baseline - 1 month - 3 months - 6 months - 12 months
  GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of sub-scales; lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100 , Higher value means better gross motor function.)
Changes in Motor Neurodevelopmental Outcome | Baseline - 1 month - 3 months - 6 months - 12 months
  Korean version of Bayley Scale of Infant Development-II Motor Scales (Higher value means better motor function: raw score 0 - worst, 112 - best)
Changes in Functional Independence in Daily Activities | Baseline - 1 month - 3 months - 6 months - 12 months
  WeeFIM (Functional Independence Measure for Children) measures functional independence in daily activities. WeeFIM contains 18 items and each item is ranked from complete dependence (scored as 1) to complete independence (scored as 7). The range is from 18 to 126 and higher scores mean more independent performance in daily activities.
Changes in Visual Perception Test | Baseline - 1 month - 3 months - 6 months - 12 months
  Visual perception function is evaluated with one of three measures: DTVP (Developmental Test of Visual Perception), MVPT (Motor-free Visual Perception Test), and VMI (Visual-Motor Integration). All can be scored as percentile rank from 0 to 100. Higher values mean better visual perception ability.
Changes in Muscle Strength | Baseline - 1 month - 3 months - 6 months - 12 months
  Summation of MMT (manual muscle testing): summated scores of the manual muscle strength test (zero=0, trace=1, poor=2, fair=3, good=4, normal=5) for flexors, extensors, abductors, and adductors of bilateral shoulder and hip joints; flexors and extensors of bilateral elbow, wrist, and knee; dorsiflexors and plantar flexors of the ankles (range: 0 ~ 160). Higher scores mean better muscle strength.
Changes in Functional Performance in Daily Activities | Baseline - 1 month - 3 months - 6 months - 12 months
  Pediatric Evaluation of Disability Inventory (PEDI) for assessing functional performance in daily activities in children (All values are adjusted and higher value means better functional performance, 0 - worst, 100 - best.)
Changes in Language Evaluation | Baseline - 6 months - 12 months
  Sequenced Language Scale for Infant (SELSI), Preschool Receptive-Expressive Language Scale (PRES) or Korean Western Aphasia Battery (K-WAB)
Changes in Brain glucose metabolism | Baseline - 12 months
  FDG-PET

CONTACTS AND LOCATIONS:
Overall Officials: MinYoung Kim, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Cha B, Kwak H, Bang JI, Jang SJ, Suh MR, Choi JI, Kim M. Safety and Efficacy of Allogeneic Umbilical Cord Blood Therapy for Global Development Delay and Intellectual Disability. Stem Cells Dev. 2023 Apr;32(7-8):170-179. doi: 10.1089/scd.2022.0252. Epub 2023 Mar 20. PMID 36734415